CLINICAL TRIAL: NCT02378220
Title: A Pilot Prospective, Randomized Controlled Trial Assessing the Clinical Impact of Integrated Pharmacogenetic Testing on Selected OASIS Metrics, Re-hospitalizations and Emergency Department Visits
Brief Title: Pharmacogenetic Testing Among Home Health Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genelex Corporation (Industry)
Collaborators: Harding University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-003
Record Dates: First submitted 2015-02-24; First posted 2015-03-04 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Adverse Drug Events; Adverse Drug Reactions; Drug Interaction Potentiation; Drug Metabolism, Poor, CYP2D6-RELATED; Drug Metabolism, Poor, CYP2C19-RELATED; Cytochrome P450 Enzyme Deficiency; Cytochrome P450 CYP2D6 Enzyme Deficiency; Cytochrome P450 CYP2C9 Enzyme Deficiency; Cytochrome P450 CYP2C19 Enzyme Deficiency; Cytochrome P450 CYP3A Enzyme Deficiency; Poor Metabolizer Due to Cytochrome P450 CYP2C9 Variant; Poor Metabolizer Due to Cytochrome p450 CYP2C19 Variant; Poor Metabolizer Due to Cytochrome P450 CYP2D6 Variant
Keywords: Home Care Agencies; Home Health Care Agencies; Home Health Care Nursing; Home Health Nurses; CYP 2D6; CYP 2C9; CYP 2C19; CYP 3A4; CYP 3A5
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Drug Metabolism, Poor, CYP2D6-Related; Drug Metabolism, Poor, CYP2C19-Related | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controls ("not tested") (No Intervention): Treatment as usual (e.g. review of potential drug-drug interactions via Lexicomp Online)
- Intervention ("tested") (Active Comparator): Patients in the "tested" group will receive pharmacogenetic testing via YouScript® Personalized Prescribing System. The study pharmacist will review drug-drug interactions (DDI), drug-gene interactions (DGI), and drug-drug-gene interactions (DDGI) using YouScript® to provide drug therapy recommendations to prescribers.
  Interventions: Genetic: Pharmacogenetic testing

INTERVENTIONS:
Genetic: Pharmacogenetic testing — Pharmacogenetic testing via YouScript® Personalized Prescribing System
  Other Names: YouScript® Personalized Prescribing System
  Arms: Intervention ("tested")

SUMMARY:
Patients meeting eligibility criteria will be randomized into two groups, one receiving pharmacogenetic testing and the other not receiving pharmacogenetic testing. In this open-label trial, a pharmacist will make medication therapy recommendations using YouScript® Personalized Prescribing System for patients who receive genetic testing and standard drug information resources per usual for patients who do not undergo pharmacogenetic testing.

DETAILED DESCRIPTION:
Both groups will be followed for 60 days. The number of re-hospitalizations and emergency department (ED) visits will be recorded as well as time to first re-hospitalization and time to first ED visit. Select Outcome and Assessment Information Set (OASIS) metrics (e.g. M1034, M1242, M1710, M1720, M1745, M2110) and Patient Health Questionnaire (PHQ)-2 will be evaluated and documented at time of admission to home health, at 30 days, and at 60 days for improvement in overall status, pain, confusion, anxiety, depression, disruptive behavior, and the need for assistance with activities of daily living (ADLs) and instrumental activities of daily living (IADLs). The number of falls will be collected as well as the proportion of YouScript® recommendations accepted by study pharmacist and passed on to clinicians and the proportion of recommendations accepted by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older.
* Willing and able to provide informed consent for study participation either directly or by a legally authorized representative (LAR).
* Presently taking or beginning treatment with at least one of the following oral forms of medication (excluding medications taken PRN) (generic name given with major U.S. brand name given in parentheses). These medications are subject to significant drug-gene interactions as defined by FDA boxed warning, FDA cautionary labeling, clinical literature or a YouScript® algorithm-predicted significant effect: Amitriptyline (Elavil), Aripiprazole (Abilify), Atomoxetine (Strattera), Carvedilol (Coreg), Celecoxib (Celebrex), Citalopram (Celexa), Clobazam (Onfi), Clomipramine (Anafranil), Clopidogrel (Plavix), Clozapine (Clozaril), Codeine [Tylenol #3 (combo)], Desipramine (Norpramin), Dextromethorphan (Delsym), Diazepam (Valium), Doxepin (Sinequan), Escitalopram (Lexapro), Esomeprazole (Nexium), Fesoterodine (Toviaz), Flecainide (Tambocor), Fluoxetine (Prozac), Flurbiprofen (Ansaid), Fluvoxamine (Luvox), Haloperidol (Haldol), Hydrocodone , Ibuprofen (Motrin), Iloperidone (Fanapt), Imipramine (Tofranil), Indomethacin (Indocin), Meloxicam (Mobic), Metoprolol (Toprol XL), Mexiletine (Mexitil), Nortriptyline (Pamelor), Omeprazole (Prilosec), Oxycodone (Oxycontin), Paroxetine (Paxil), Perphenazine (Trilafon), Phenobarbital (Luminal), Phenytoin (Dilantin), Pimozide (Orap), Piroxicam (Feldene), Proguanil [(Malarone (combo)], Propafenone (Rythmol), Propranolol (Inderal), Risperidone (Risperdal), Sertraline (Zoloft), Tetrabenazine (Xenazine), Thioridazine (Mellaril), Timolol (Apotimol), Tolterodine (Detrol), Torsemide (Demadex), Tramadol (Ultram), Trimipramine (Surmontil), Venlafaxine (Effexor), Voriconazole (Vfend), Vortioxetine (Brintellix), Warfarin (Coumadin).

Exclusion Criteria:

* Previous CYP testing (CPT codes 81225, 81226, 81227, 81355, 81401)
* History of organ transplant (199.2; 238.77; 414.06; 414.07; 996.80-996.89; E878.0; V42.0-V42.7; V42.81-V42.84; V42.89; V42.9; V45.87; V49.83; V58.44)
* Current malabsorption syndrome (579.0), including the following: Intestinal malabsorption (579.8, 579.9), Postoperative malabsorption (579.3), or Short bowel syndrome (579.3)
* Treatment of invasive solid tumors or hematologic malignancies in the last year, excluding in situ cancers or non-melanoma skin cancer (basal cell carcinoma)
* End Stage Renal Disease (ESRD)
* Persistent acute renal failure: complete loss of kidney function >4 weeks (requiring dialysis)
* Renal failure by: Glomerular filtration rater (GFR): SCr > 3 times baseline or GFR decreased 75% or SCr ≥4 mg/dL; acute rise ≥0.5 mg/dL; OR Urine Output (UO): UO < 0.3 mL/kg/h 24 h (oliguria) or anuria 12 h.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Elliott, PharmD, Principal Investigator — Harding University
Locations (1):
- White County Medical Center Home Health, Searcy, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Elliott LS, Henderson JC, Neradilek MB, Moyer NA, Ashcraft KC, Thirumaran RK. Clinical impact of pharmacogenetic profiling with a clinical decision support tool in polypharmacy home health patients: A prospective pilot randomized controlled trial. PLoS One. 2017 Feb 2;12(2):e0170905. doi: 10.1371/journal.pone.0170905. eCollection 2017. PMID 28151991
- See also: Clinical impact of pharmacogenetic profiling with a clinical decision support tool in polypharmacy home health patients: A prospective pilot randomized controlled trial — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0170905
- See also: PGx Testing Firm Genelex Publishes RCT, Spins Out Analytics Unit in Effort to Improve Adoption — https://www.genomeweb.com/molecular-diagnostics/pgx-testing-firm-genelex-publishes-rct-spins-out-analytics-unit-effort-improve
- See also: Genomics, Clinical Decision Support Combo Cuts ED Visits by 42% — http://healthitanalytics.com/news/genomics-clinical-decision-support-combo-cuts-ed-visits-by-42

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at a hospital-based HHA in Searcy, Arkansas. The study population was derived from patient referrals to home health upon hospital discharge. Of 655 patients assessed for eligibility, 412 did not meet the inclusion criteria and 133 patients declined to participate.
Pre-assignment Details: Exclusion criteria were the same for tested and untested groups and included patients previously tested for CYP 450, history of organ transplant, current malabsorption, treatment of invasive solid tumors or hematologic malignancies in the last year, end stage renal disease or current dialysis.
Groups:
- Intervention ("Tested"): Patients in the "tested" group will receive pharmacogenetic testing via YouScript® Personalized Prescribing System. The study pharmacist will review drug-drug, drug-gene, and drug-drug-gene interactions using YouScript® to provide drug therapy recommendations to prescribers.
  Pharmacogenetic testing: Pharmacogenetic testing via YouScript® Personalized Prescribing System
Period: Overall Study
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Started (Patients were enrolled from Feb 2015 to Dec 2015 with follow-up ending in Feb 2016.) | 53 | 57
Completed | 47 | 56
Not Completed | 6 | 1
Not completed — Death | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls ("Not Tested") | Intervention ("Tested") | Total
Number analyzed (Participants) | 53 | 57 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 39 | 51 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline data was extracted from patient charts & manually entered into the study database.Study pharmacist reviewed DDIs, DGIs, and cumulative drug and/or gene interactions in the tested group using the YouScript generated reports and CDST to provide drug therapy recommendations to clinicians, after which prescriptions were altered at clinician discretion. Patients in the untested group were screened for DDIs using standard drug information resources (Lexicomp) with recommendations acted on according to clinician judgment. Time to change therapy was similar to those in the tested group.
  years | 74.6 (11.9) | 76.5 (9.4) | 75.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 17 | 25 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 52 | 57 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 57 | 110
OASIS Metrics [Mean (Full Range); unit: Scores on a scale] — OASIS (Outcome and Assessment Information Set) Score represents an outcome measure in home health at an individual patient level to plan care, measure quality, and calculate reimbursement. On an overall scale of 0 to 3, a lower number represents a better outcome.
  Average Pharmacogenetic Risk score estimates individual patient risk of having at least one significant adverse drug event due to genetic variation. Total range is 0 to 100, representing percentage, where a larger number indicates a higher risk.
  Scores on a scale
    OVERALL OASIS SCORE | 1.63 [0 to 3] | 1.64 [0 to 3] | 1.63 [0 to 3]
    AVERAGE PHARMACOGENETIC RISK | 34.3 [0 to 73] | 33.2 [0 to 63] | 33.75 [0 to 73]

OUTCOME MEASURES:

1. Primary Outcome: Number of Re-hospitalizations at 30 and 60 Days
Description: The primary outcomes included the number of re-hospitalizations at 30 and 60 days.
Time Frame: 30 days, 60 days post discharge
Population: Primary outcomes included the number of re-hospitalizations between the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Re-hospitalizations
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Re-hospitalizations
  Re-hospitalizations at 30 Days | 0.38 [0 to 2] | 0.25 [0 to 3]
  Re-hospitalizations at 60 Days | 0.7 [0 to 3] | 0.33 [0 to 3]
Statistical Analysis 1: Comparison: Controls ("Not Tested") vs Intervention ("Tested"); Test type: Other; p = 0.21, Regression, Poisson — P-value for 30 days measure; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.32 to 1.28]
Statistical Analysis 2: Comparison: Controls ("Not Tested") vs Intervention ("Tested"); Test type: Other; p = 0.007, Regression, Poisson — P-Value for 60 days measure; Risk Ratio (RR) = 0.48, 95% CI 2-sided [0.27 to 0.82]

2. Primary Outcome: The Primary Outcomes Included the Number of Emergency Department Visits at 30 and 60 Days.
Description: Assessed the number of Emergency Department visits at 30 and 60 days post discharge with pharmacogenetic testing and YouScript® Personalized Prescribing system.
Time Frame: 30 days, 60 days post discharge
Population: The primary outcomes assessed the number of emergency department visits between the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: ED visits
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
ED visits
  ED Visits at 30 Days | 0.40 [0 to 2] | 0.25 [0 to 2]
  ED Visits at 60 Days | 0.66 [0 to 4] | 0.39 [0 to 2]
Statistical Analysis 1: Comparison: Controls ("Not Tested") vs Intervention ("Tested"); Test type: Other; p = 0.16, Regression, Poisson — P-Value for 30 days measure; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.31 to 1.21]
Statistical Analysis 2: Comparison: Controls ("Not Tested") vs Intervention ("Tested"); Test type: Other; p = 0.045, Regression, Poisson; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.34 to 0.99]

3. Secondary Outcome: Time to 1st Re-hospitalization
Description: To assess time to first re-hospitalization, we compared the exploratory time-to-event outcomes between the tested and untested groups at 30 days and 60 days. These outcomes were measured using cumulative percentage events at 30 and 60 days, referring to the percentage of subjects re-hospitalized before or at 30 and 60 days.
Time Frame: 30 days, 60 days
Population: We compared the exploratory time-to-event outcomes between the tested and untested groups at 30 days and 60 days.
Measure: Number; unit: Percentage of participants
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Percentage of participants
  Cumulative Percentage Events at 30 Days | 29 | 19
  Cumulative Percentage Events at 60 Days | 43 | 28
Statistical Analysis 1: Comparison: Controls ("Not Tested") vs Intervention ("Tested"); Test type: Other; p = 0.10, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.31 to 1.12]

4. Secondary Outcome: Time to 1st Emergency Department Visit
Description: To assess time to first emergency department visit, we compared the exploratory time-to-event outcomes (time to 1st ED visit) between the tested and untested groups at 30 days and 60 days. These outcomes were measured using cumulative percentage events at 30 and 60 days, referring to the percentage of subjects who visited the emergency department before or at 30 and 60 days.
Time Frame: 30 days, 60 days
Population: Compared the exploratory time-to-event outcomes between the tested and untested groups at 30 days and 60 days.
Measure: Number; unit: Percentage of participants
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Percentage of participants
  Cumulative Percentage Events at 30 Days | 30 | 23
  Cumulative Percentage Events at 60 Days | 49 | 32
Statistical Analysis 1: Comparison: Controls ("Not Tested") vs Intervention ("Tested"); Test type: Other; p = 0.09, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.33 to 1.10]

5. Secondary Outcome: Overall Status as Measured by Outcome and Assessment Information Set (OASIS) Scale
Description: We assessed the impact of genetic testing on overall status according to OASIS M1034 at 30 and 60 days post discharge. OASIS measures various data items to assess home health care quality and performance. OASIS M1034, one data point in the OASIS system, measures overall patient status on a scale of 0 to 3, with a lower score indicating better overall status.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed the overall status according to OASIS M1034 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS M1034 at 30 Days | 1.00 [0 to 2] | 1.11 [0 to 3]
  OASIS M1034 at 60 Days | 0.76 [0 to 3] | 0.71 [0 to 3]

6. Secondary Outcome: Pain as Measured by OASIS Scale
Description: We assessed the impact of genetic testing on patient pain frequency according to OASIS M1242 at 30 and 60 days post discharge. OASIS measures various data items to assess home health care quality and performance. OASIS M1242, one data point in the OASIS system, measures patient pain frequency on a scale of 0 to 4, with a lower score indicating less frequent pain.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed frequency of pain according to OASIS M1242 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS M1242 at 30 Days | 1.02 [0 to 4] | 1.16 [0 to 4]
  OASIS M1242 at 60 Days | 1.19 [0 to 4] | 1.49 [0 to 4]

7. Secondary Outcome: Confusion as Measured by OASIS Scale
Description: We assessed the impact of genetic testing on frequency of confusion according to OASIS M1710 at 30 and 60 days post discharge. OASIS measures various data items to assess home health care quality and performance. OASIS M1710, one data point in the OASIS system, measures patient confusion frequency on a scale of 0 to 4, with a lower score indicating less frequent confusion.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed frequency of confusion according to OASIS M1710 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS M1710 at 30 Days | 0.49 [0 to 4] | 0.66 [0 to 3]
  OASIS M1710 at 60 Days | 0.79 [0 to 4] | 0.61 [0 to 4]

8. Secondary Outcome: Anxiety as Measured by OASIS Scale
Description: We assessed the impact of genetic testing on frequency of anxiety according to OASIS M1720 at 30 and 60 days post discharge. OASIS measures various data items to assess home health care quality and performance. OASIS M1720, one data point in the OASIS system, measures patient confusion frequency on a scale of 0 to 3, with a lower score indicating less frequent confusion.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed frequency of anxiety according to OASIS M1720 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS M1720 at 30 Days | 0.51 [0 to 3] | 0.41 [0 to 2]
  OASIS M1720 at 60 Days | 0.67 [0 to 3] | 0.55 [0 to 2]

9. Secondary Outcome: Depression as Measured by Patient Health Questionnaire (PHQ)-2 Scale
Description: We assessed the impact of genetic testing on frequency of depressive mood according to PHQ-2 at 30 and 60 days post discharge. PHQ-2 evaluates patient depression by assessing two factors: frequency of little interest or pleasure in doing things and frequency of feeling down, depressed, or hopeless. This outcome measure assessed the second factor, frequency of feeling down or depressed. The scale for this factor ranges from 0 to 3, with a lower score represented less frequent depressive feelings.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed feelings of depression according to PHQ-2 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS PHQ-2 at 30 Days | 0.06 [0 to 1] | 0.16 [0 to 2]
  OASIS PHQ-2 at 60 Days | 0.59 [0 to 3] | 0.35 [0 to 2]

10. Secondary Outcome: Disruptive Behavior as Measured by OASIS Scale
Description: We assessed the impact of genetic testing on frequency of disruptive behavior according to OASIS M1745 at 30 and 60 days post discharge. OASIS measures various data items to assess home health care quality and performance. OASIS M1745, one data point in the OASIS system, measures frequency of disruptive behavior by patient on a scale of 0 to 5, with a lower score indicating less frequent disruptive behavior.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed frequency of disruptive behavior according to OASIS M1745 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS M1745 at 30 Days | 0.06 [0 to 1] | 0.05 [0 to 1]
  OASIS M1745 at 60 Days | 0.45 [0 to 5] | 0.14 [0 to 3]

11. Secondary Outcome: Activities of Daily Living as Measured by OASIS Scale
Description: We assessed the impact of genetic testing on the frequency of activities of daily living (ADL) and instrumental activities of daily living (IADL) assistance according to OASIS M2110 at 30 and 60 days post discharge. OASIS measures various data items to assess home health care quality and performance. OASIS M2110, one data point in the OASIS system, measures frequency of receiving ADL/IADL assistance on a scale of 0 to 5, with a lower score indicating less frequent assistance.
Time Frame: 30 days, 60 days post discharge
Population: The secondary outcomes assessed frequency of ADL and IADL according to OASIS M2110 of the tested group and the untested group at 30 and 60 days post-discharge.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Scores on a scale
  OASIS M2110 at 30 Days | 2.72 [1 to 5] | 2.30 [1 to 5]
  OASIS M2110 at 60 Days | 2.86 [1 to 5] | 2.76 [1 to 5]

12. Secondary Outcome: Number of Falls as Measured by Tabulation
Description: To assess whether YouScript® testing decreases falls
Time Frame: 60 days
Measure: Mean (Full Range); unit: Falls
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
Number analyzed (Participants) | 53 | 57
Falls | 0.09 [0 to 1] | 0.11 [0 to 1]

13. Secondary Outcome: Number of Pharmacist-accepted of Recommendations as Measured by Tabulation
Description: To assess the proportion of YouScript® Personalized Prescribing System recommendations accepted by the study pharmacist and passed on to clinicians.
Time Frame: 60 days
Population: This secondary outcome assessed the proportion of YouScript® Personalized Prescribing System recommendations provided for patients in the "tested" group accepted by the study pharmacist and passed to clinicians.
Measure: Number; unit: recommendations
Arm/Group | Intervention ("Tested")
Number analyzed (Participants) | 57
recommendations
  Number of YouScript® Recommendations Made | 124
  Number of YouScript® Recommendations Accepted | 124

14. Secondary Outcome: Number of Clinician-accepted of Recommendations as Measured by Tabulation
Description: To assess the proportion of study pharmacist recommendations acted on by clinicians.
Time Frame: 60 days
Population: This secondary outcome assessed the proportion of YouScript® Personalized Prescribing System recommendations provided for patients in the "tested" group acted on by clinicians.
Measure: Number; unit: recommendations
Arm/Group | Intervention ("Tested")
Number analyzed (Participants) | 57
recommendations
  Number of Recommendations Passed to Clinicians | 124
  Number of Recommendations Followed | 96
  Number of Recommendations Not Followed | 6
  Number of Unknown Status Recommendations | 22

ADVERSE EVENTS:
Time Frame: We compared primary and exploratory composite outcomes (re-hospitalizations, ED visits and mortality) between the tested group and the untested group at 30 and 60 days post-discharge. The adverse events were not recorded.
Description: The adverse events were not tracked and was not an outcome of our study. However, we compared differences in the distribution of CYP 450 metabolic phenotypes, and differences in the severity of drug-drug interactions (DDI) (binary and cumulative), drug-gene interactions (DGI), or drug-drug-gene interactions (DDGI) between this home health trial and another published study population.
Arm/Group | Controls ("Not Tested") | Intervention ("Tested")
All-Cause Mortality (participants affected / at risk) | 6/53 | 1/57
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The limitations of this study include small sample size, use of a randomized population within one institution and undetermined impact of the genetic testing on patient-provider interactions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No